CLINICAL TRIAL: NCT03450876
Title: A Prospective Multicenter Cohort Study of Late Physical Psychological and Social Effects in Patients Treated With Ipilimumab for Advanced Melanoma
Brief Title: Long Term Quality of Life in Melanoma Patients in Netherlands
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-483
Record Dates: First submitted 2018-02-15; First posted 2018-03-01 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Healthy Control: Individuals without melanoma (stage III or IV) diagnosis that have been included in the PROFILES cohort
  Interventions: Other: Non-Interventional
- 24 to < 36 months post-ipilimumab treatment: 24 to 36 month post-ipilimumab treatment advanced melanoma patients that were treated with ipilimumab in 2014 in one of the 14 melanoma centers in the Netherlands
  Interventions: Other: Non-Interventional
- ≥ 36 to < 48 months post-ipilimumab treatment: 36 to 48 month post-ipilimumab treatment advanced melanoma patients that were treated with ipilimumab in 2013 in one of the 14 melanoma centers in the Netherlands
  Interventions: Other: Non-Interventional
- ≥ 48 months post-ipilimumab treatment: Greater than 48 month post-ipilimumab treatment advanced melanoma patients that were treated with ipilimumab between 2011 and 2012 in one of the 14 melanoma centers in the Netherlands
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
Study of late physical, psychological and social effects in patients treated with ipilimumab for advanced (stage IV or unresectable stage III) melanoma.

ELIGIBILITY:
Inclusion Criteria-

* Patient population: Adults ≥ 18 years of age at diagnosis, diagnosed with histologically confirmed advanced (stage IV or unresectable stage III) melanoma, who have received at least one course of ipilimumab treatment (first, second, or second plus line; routine practice or study treatment) in one of the specified treatment centers, and who have survived at least 2 years after (completion of) ipilimumab treatment (measured from last ipilimumab administration)
* Matched healthy control population: Individuals without melanoma (stage III or IV) diagnosis that have been included in the PROFILES cohort

Exclusion Criteria

* Insufficient understanding of the Dutch language
* Other anticancer treatment after ipilimumab or during study entry
* Disease recurrence during the study

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with advanced melanoma who survived at least 2 years and were treated with ipilimumab between 2011 and 2015 in one of the specified melanoma centers in the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
European Organisation for Research and Treatment of Cancer Quality of Life questionnaire (EORTC QLQ C30) | Baseline up to 3 years
  EORTC QLQ-C30 is a self-reported, 30-item generic questionnaire developed to assess 15 domains: global health status scale, five functional scales (physical, role, emotional, cognitive, and social functioning) and nine symptom scales (fatigue, nausea, vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties).

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Baseline up to 3 years
  14-item questionnaire assesses symptoms of mood disturbance, yielding separate scale scores for anxiety and depression, as well as a total score
Multidimensional Fatigue Inventory (MFI) | Baseline up to 3 years
  Fatigue will be assessed with the Multidimensional Fatigue Inventory (MFI)
Cancer Worry Scale (CWS) | Baseline up to 3 years
  8-item questionnaire will be used to assess the prevalence of cancer-specific distress in melanoma survivors and in healthy controls
European Organisation for Research and Treatment of Cancer Quality Of Life (EORTC QLQ) module for sexual health | Baseline up to 3 years
  Sexual health will be assessed with the European Organisation for Research and Treatment of Cancer Quality Of Life (EORTC QLQ) module for sexual health
Functional Assessment of Cancer Therapy-Melanoma questionnaire (FACT-M) | Baseline up to 3 years
  51-item measurement of quality of life
EuroQOL-5D (EQ-5D) survivors | Baseline up to 3 years
  Generic health status will be assessed with the EuroQOL-5D (EQ-5D) survivors
Impact of Cancer Questionnaire (IOCv2) | Baseline up to 3 years
  81 items that present statements regarding specific impacts of cancer to which respondents indicate their level of agreement from 1 (strongly disagree) to 5 (strongly agree). Seventy items apply to all survivors, 3 to currently employed respondents, 4 to respondents not currently partnered, and 4 to currently partnered respondents
Work Ability Index questionnaire (WAI) | Baseline up to 3 years
  13-item questionnaire developed to obtain survivors' experiences with return to work and work performance
EORTC information module (EORTC QLQINFO25) | Baseline up to 3 years
  Information needs will be assessed with the EORTC information module (EORTC QLQINFO25)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Amsterdam, Netherlands

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm